CLINICAL TRIAL: NCT00311740
Title: A Multi-center, Factorial Study to Evaluate Efficacy & Safety of 8 Wks Treatment With VAH631 [Valsartan (40 & 80 mg) and Hydrochlorothiazide (6.25 & 12.5 mg) Combined & Alone in Essential Hypertensive Patients] - Double-blind Study of VAH631 in Patients With Essential Hypertension (Factorial Study)
Brief Title: A Study of VAH631 in Patients With Essential Hypertension (Factorial Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: CVAH631B1303
Record Dates: First submitted 2006-04-04; First posted 2006-04-06 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Hypertension
Keywords: Hypertension,; Valsartan,; Hydrochlorothiazide
MeSH Terms: conditions — Hypertension | interventions — Valsartan; Hydrochlorothiazide

INTERVENTIONS:
Drug: Valsartan
Drug: Hydrochlorothiazide

SUMMARY:
The purpose of this study is to compare the effect of the fixed combination of valsartan+hydrochlorothiazide (HCTZ) on blood pressure reduction with valsartan and HCTZ alone and whether the combination treatments are safe and well tolerated. The study aims to establish a dose response relationship for both monotherapies and the combinations.

This study is being conducted in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Essential hypertension measured by mercury sphygmomanometer
* Outpatients

Exclusion Criteria:

* Secondary hypertension or suspected of having secondary hypertension.
* A history of malignant hypertension
* Severe hypertension
* Significant heart, renal, hepatic diseases or significant cerebrovascular disorder
* Gout Other protocol-defined inclusion/exclusion criteria may apply

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 582 (Actual)
Dates: Start 2006-03; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in diastolic blood pressure after 8 weeks

SECONDARY OUTCOMES:
Change from baseline in systolic blood pressure after 8 weeks
Diastolic blood pressure less than 90 mmHg or at least a 10 mmHg decrease in diastolic blood pressure after 8 weeks
Change from baseline in standing diastolic blood pressure after 8 weeks
Change from baseline in standing systolic blood pressure after 8 weeks
Adverse events and serious adverse events at each study visit for 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novatis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, Tokyo, Japan